CLINICAL TRIAL: NCT06217094
Title: Phase I Study of NP-101 in Patients With Unresectable Hepatocellular Carcinoma (HCC) Undergoing Y-90 Treatment
Brief Title: Study of NP-101 in Patients With Unresectable Hepatocellular Carcinoma (HCC) Undergoing Y-90 Treatment
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: insufficient staff
Sponsor: University of Florida (Other)
Collaborators: Novatek (Unknown); Florida Department of Health (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: UF-GI-018; OCR44171 (Other: University of Florida); IRB202401248 (Other: University of Florida)
Record Dates: First submitted 2024-01-10; First posted 2024-01-22 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; NP-101; Y-90
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- NP-101 (3 g) (Experimental)
  Interventions: Drug: NP-101 (3 g)
- NP-101 (4.8 g) (Experimental)
  Interventions: Drug: NP-101 (4.8 g)
- NP-101 (6 g) (Experimental)
  Interventions: Drug: NP-101 (6 g)

INTERVENTIONS:
Drug: NP-101 (3 g) — Subjects will be assigned to take 3 g of NP-101 orally once daily for 28 days pre Y-90 treatment.
  Arms: NP-101 (3 g)
Drug: NP-101 (4.8 g) — Subjects will be assigned to take 4.8 g of NP-101 orally once daily for 28 days pre Y-90 treatment.
  Arms: NP-101 (4.8 g)
Drug: NP-101 (6 g) — Subjects will be assigned to take 6 g of NP-101 orally once daily for 28 days pre Y-90 treatment.
  Arms: NP-101 (6 g)

SUMMARY:
Surgical resection and liver transplantation are the primary curative treatments for hepatocellular carcinoma (HCC). However, many patients are ineligible for these treatments due to advanced disease, social factors, or limited availability of liver donors. Therefore, for patients with unresectable HCC, locoregional therapies like transarterial radioembolization (TARE with Y90) are considered the next best non-operative option, especially when the cancer remains confined to the liver. Despite the use of these liver-directed therapies, relapse rates and mortality remain high, underscoring the need for new predictive biomarkers and therapeutic targets, including immune modulation.

The rationale behind NP-101 (TQ formula) stems from its immune modulatory properties as a potent drug derived from a natural substance, black seed or Nigella Sativa. Previous studies have demonstrated its immune modulation and anti-cancer effects, showing promise in preclinical models of HCC. In a randomized phase 2 study conducted in Covid patients, NP-101 exhibited safety and significantly increased T effector cells (CD4+ and CD8+ T lymphocytes), resulting in accelerated recovery. The immune modulation effect of NP-101, observed in the Covid study, and its potential to enhance CD4+ and CD8+ T effector lymphocytes can potentially modify the immune microenvironment and improve outcomes in locally advanced HCC patients undergoing Y90 treatment.

This study will investigate the safety, efficacy and maximum tolerated dose of NP-101 in patients with unresectable hepatocellular carcinoma.

The dosing scheme for NP-101 in this study will follow a Bayesian Optimal Interval design. Based on the target dose-limiting toxicity (DLT) rate of 30% and assuming a 3+3 design, three subjects will be sequentially enrolled at each of the 3 dose levels (beginning with 3g) until at least one DLT occurs.

If no DLTs occur, dosing will be escalated to the next dose level for the next three enrolled subjects. At either of the two dose levels, if 1 DLT occurs, three more subjects will be enrolled at that dose level. If no DLTs occur in these subjects, three more subjects will be enrolled at the next highest dose level. Dosing escalation will be stopped if two or more total DLTs occur at any dose level. The maximum tolerated dose (MTD) will be one dose level below the dose level at which two or more DLTs occurred.

ELIGIBILITY:
Inclusion Criteria:

* Must provide written informed consent prior to initiating any trial related procedures
* Adults ≥ 18 years of age
* Patient has histologically or radiographically confirmed HCC. Initial HCC diagnosis during study screening can also be made based on characteristic imaging pattern per the AASLD (American Association for the Study of Liver Diseases) guidelines (https://journals.lww.com/hep/fulltext/2023/12000/aasld_practice_guidance_on_prevention,_diagnosis,.27.aspx). Per AASLD guidelines: "arterial phase hyperenhancement (APHE) and washout on portal venous or delayed phases of contrast-enhanced multiphase CT or MRI are considered radiological hallmarks of HCC given high specificity and positive predictive value in lesions ≥1 cm in size."
* Unresectable HCC or not eligible for surgical resection or liver transplantation at the time of screening.
* At least one untreated target lesion that could be measured in one dimension, according to the modified Response Evaluation Criteria in Solid Tumors (mRECIST).
* Must have a Child-Turcotte-Pugh score of Class A (5-6) or B7
* ECOG of 0 or 1
* Adequate hematologic, renal, and coagulation function, as evidenced by:

  * Hemoglobin ≥ 9 g/dL
  * Absolute neutrophil count ≥ 1,500/mm3
  * Platelet count ≥ 75,000/mm3
  * Creatinine clearance ≥ 30 mL/min
  * International Normalized Ratio (INR) ≤ 1.5 or prothrombin time ≤ 3 seconds above control
  * Total bilirubin level of ≤ 2.0 mg/dL
* Subjects of childbearing potential (SOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for at least 12 weeks after the last dose of study drug to minimize the risk of pregnancy. Prior to study enrollment, subjects of childbearing potential must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy.
* Subjects with partners of child-bearing potential must agree to use physician-approved contraceptive methods (e.g., abstinence, condoms, vasectomy) throughout the study and should avoid conceiving children for 12 weeks following the last dose of study drug.

Exclusion Criteria:

* Patient has been treated for this malignancy, has another active malignancy, or has had an active malignancy within the last two years.
* Previous treatment with Y90 radioembolization or systemic treatment for HCC.
* Evidence of macrovascular invasion or extrahepatic metastases.
* Patient has fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC where HCC is not the majority histology.
* Patients who experienced recent GI bleeding or intracranial bleeding or stroke in last 12 weeks, or with uncontrolled blood pressure of history of organ rupture or perforation in last 12 weeks.
* Prior liver transplantation.
* Subjects of childbearing potential who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for at least 12 weeks after the last dose of study drug.
* Subjects who are confirmed to be pregnant or breastfeeding.
* History of any other disease, metabolic dysfunction, clinical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of protocol therapy or that might affect the interpretation of the results of the study or that puts the subject at high risk for treatment complications, in the opinion of the treating physician.
* Administration of a vaccine containing live virus within 30 days prior to the first dose of trial treatment. Note: Most flu vaccines are killed viruses, with the exception of the intra-nasal vainer (Flu-Mist) which is an attenuated live virus and therefore prohibited for 30 days prior to first dose. Non-live versions of the COVID vaccine are allowed.
* Prisoners or subjects who are involuntarily incarcerated, or subjects who are compulsorily detained for treatment of either a psychiatric or physical illness
* Use of immunosuppressive drugs, such as steroids, and any herbs, which cannot be discontinued prior to study entry

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose | 2 months
  Determine the maximum tolerated dose of NP-101

SECONDARY OUTCOMES:
Overall response rate | 20 weeks
  Determine the overall response rate. Overall response rate is defined as the percentage of participants who have a confirmed complete response or partial response, as determined by mRECIST.
Disease control rate | 20 weeks
  Determine the disease control rate, which is defined as the percentage of participants who have experienced either a complete response, a partial response, or stable disease per mRECIST criteria.
Duration of response | 20 weeks
  Determine the duration of response, which is defined as the the time from the date of first documented response until the date of documented progression per mRECIST or death due to any cause.
Progression-free survival | 1 year
  Determine the progression-free survival, which is defined as time between first study treatment and first documentation of disease progression using RECIST criteria, or to death due to any cause, whichever comes first.
Overall survival | 172 weeks
  Determine the overall survival, which is defined as time between first study treatment and the date of death due to any cause. In the absence of confirmation of death, survival time will be censored at the last date the subject is known to be alive.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Zarrinpar, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States